CLINICAL TRIAL: NCT06949657
Title: Occurrence and Influencing Factors of Cognitive Impairment in Elderly Patients With Schizophrenia and the Application Effect of Acceptance and Commitment Therapy Nursing Model
Brief Title: Occurrence and Influencing Factors of Cognitive Impairment in Elderly Patients With Schizophrenia and
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the sponsor has determined that access to the full dataset is no longer available
Sponsor: Third People's Hospital, Huzhou City, Zhejiang Province, China (Other)
Responsible Party: Principal Investigator, Ying Xu, Principal Investigator, Third People's Hospital, Huzhou City, Zhejiang Province, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: No. 2025-130
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia Disorders; Cognitive Impairment; Acceptance and Commitment Therapy
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the conventional treatment group (Other): Patients received conventional mental health education once weekly for 6 weeks, covering schizophrenia symptoms, treatment, and prognosis. Standard nursing care and antipsychotic medications (e.g., olanzapine, quetiapine) were maintained without additional psychological interventions.
  Interventions: Other: the conventional treatment group
- the ACT group (Other): Patients received ACT-based nursing interventions tailored to risk factors (e.g., age ≥70, long disease duration), including:
  ACT modules: Acceptance, cognitive defusion, mindfulness, values clarification, and committed action.
  Adjunct strategies: Family therapy, Tai Chi, and crisis planning. Frequency: Daily practice + 1-2 group sessions/week for 6 weeks. Goal: Enhance psychological flexibility, reduce stigma, and improve cognitive function.
  Interventions: Other: the ACT group

INTERVENTIONS:
Other: the conventional treatment group — Patients received conventional mental health education once weekly for 6 weeks, covering schizophrenia symptoms, treatment, and prognosis. Standard nursing care and antipsychotic medications (e.g., olanzapine, quetiapine) were maintained without additional psychological interventions.
  Arms: the conventional treatment group
Other: the ACT group — Patients received ACT-based nursing interventions tailored to risk factors (e.g., age ≥70, long disease duration), including:
  ACT modules: Acceptance, cognitive defusion, mindfulness, values clarification, and committed action.
  Adjunct strategies: Family therapy, Tai Chi, and crisis planning. Frequency: Daily practice + 1-2 group sessions/week for 6 weeks. Goal: Enhance psychological flexibility, reduce stigma, and improve cognitive function.
  Arms: the ACT group

SUMMARY:
ACT combined with stratified intervention improved cognitive function and quality of life in elderly schizophrenia patients by enhancing psychological flexibility and family support.

DETAILED DESCRIPTION:
This study analyzes factors influencing cognitive impairment and evaluates the efficacy of a stratified intervention combining Acceptance and Commitment Therapy (ACT) with these factors to improve cognitive function and quality of life. A total of 149 elderly patients with schizophrenia were enrolled, split into cognitive impairment (n = 86) and non-cognitive impairment (n = 63) groups. A combined case-control and randomized controlled trial design was employed. Logistic regression was used to identify independent risk factors. Cognitive impairment patients were randomly assigned to either the conventional treatment group (n = 39) or the ACT group (n = 39) for a 6-week intervention. Evaluation instruments included the AAQ-II (psychological flexibility), GSES (self-efficacy), FACES II-CV (family functioning), SSMI-C (internalized stigma), and SQLS (quality of life).

ELIGIBILITY:
Inclusion Criteria:

* (1)Meets the diagnostic criteria for schizophrenia as defined in the International Classification of Diseases, Tenth Revision (ICD-10);
* (2) age > 60 years;
* (3)possesses at least a primary school education, enabling independent completion of all questionnaires;
* (4) has been taking antipsychotic medication continuously and regularly for at least one year during the enrollment period, with current symptoms and disease status stabilized in the maintenance phase;
* (5)informed consent obtained from the patient or their family/guardian.

Exclusion Criteria:

* (1) Coexisting organic mental disorders, affective disorders, or similar conditions;
* (2) coexisting physical illnesses that may affect cognitive function, such as hepatic or renal dysfunction;
* (3) alcohol dependence or dependence on psychoactive substances;
* (4) receipt of electroconvulsive therapy within the past three months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Function | Baseline to 6 weeks post-intervention
  Improvement in global cognitive function assessed via the Montreal Cognitive Assessment (MoCA), focusing on memory, attention, and executive function. Higher scores indicate better cognition (range: 0-30).

SECONDARY OUTCOMES:
Psychological Flexibility (AAQ-II) | Baseline to 6 weeks.
  Scores on the Acceptance and Action Questionnaire-II (7 items, Likert scale 1-7). Lower scores indicate greater flexibility.
Self-Efficacy (GSES) | Baseline to 6 weeks.
  General Self-Efficacy Scale (10 items, scores 10-40). Higher scores reflect stronger self-efficacy.
Family Functioning (FACES II-CV) | Baseline to 6 weeks.
  Family Adaptability and Cohesion Evaluation Scale (cohesion + adaptability subscales). Higher scores indicate healthier family dynamics.
Stigma Reduction (SSMI-C) | Baseline to 6 weeks.
  Stigma Scale for Mental Illness (28 items). Lower scores on Discrimination/Illness Concealment subscales indicate reduced stigma.
Quality of Life (SQLS) | Baseline to 6 weeks.
  Schizophrenia Quality of Life Scale (30 items). Lower scores indicate better QoL in psychosocial, motivation, and symptom domains.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Xu, Principal Investigator — Huzhou Third People's Hospital
Locations (1):
- Huzhou Third People's Hospital, Huzhou, China